CLINICAL TRIAL: NCT00716027
Title: Applying Social Comparison Theory to Behavioral Weight Loss: Does Modifying Group Membership Improve Outcome?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Miriam Hospital (Other)
Responsible Party: Rena R. Wing, PhD, The Miriam Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2034-08
Record Dates: First submitted 2008-07-15; First posted 2008-07-16 (Estimated); Last update posted 2010-09-29 (Estimated); Status verified 2008-07

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): A 24-week intervention in which individuals will meet weekly to be instructed on behavioral change associated with weight loss, including modifying dietary intake, self-monitoring weight and eating behaviors, and increasing physical activity.
  Interventions: Behavioral: Standard behavioral treatment for weight loss
- 2 (Experimental): A 24-week intervention in which individuals will meet weekly to be instructed on behavioral change associated with weight loss, including modifying dietary intake, self-monitoring weight and eating behaviors, and increasing physical activity. In this intervention, individuals not meeting weight loss goals will be given one-on-one treatment.
  Interventions: Behavioral: Modified behavioral treatment for weight loss

INTERVENTIONS:
Behavioral: Standard behavioral treatment for weight loss — A 24-week intervention in which individuals will meet weekly to be instructed on behavioral change associated with weight loss, including modifying dietary intake, self-monitoring weight and eating behaviors, and increasing physical activity.
  Arms: 1
Behavioral: Modified behavioral treatment for weight loss — A 24-week intervention in which individuals will meet weekly to be instructed on behavioral change associated with weight loss, including modifying dietary intake, self-monitoring weight and eating behaviors, and increasing physical activity. In this intervention, individuals not meeting weight loss goals will be given one-on-one treatment.
  Arms: 2

SUMMARY:
The purpose of this study is to determine whether a modified behavioral treatment for weight loss that includes one-on-one treatment for individuals struggling to lose weight is associated with more weight loss than a standard behavioral treatment.

ELIGIBILITY:
Inclusion Criteria:

* BMI between 27 and 45 kg/m2

Exclusion Criteria:

* participating in a weight loss program or taking a weight loss medication
* currently pregnant, lactating, or less than 6-months post-partum or plan to become pregnant during the time of the intervention.
* report a heart condition, chest pain during periods of activity or rest, or loss of consciousness
* report conditions that would render the participant unlikely to follow the study protocol (e.g., terminal illness, relocation, substance abuse, sever psychiatric condition, dementia).

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2008-07; Primary Completion 2009-12 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
weight | weekly for 24-weeks

CONTACTS AND LOCATIONS:
Overall Officials: Rena R Wing, PhD, Principal Investigator — The Miriam Hospital
Locations (1):
- The Miriam Hospital, Providence, Rhode Island, United States